CLINICAL TRIAL: NCT07204522
Title: Observational Study on the Efficacy of Empirical Antimicrobial Therapy in Febrile Neutropenia.
Brief Title: Efficacy of Empirical Anti-Infective Therapy in Neutropenic Febrile Patients.
Status: Recruiting | Type: Observational
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanxiBethuneH3
Record Dates: First submitted 2025-09-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia | interventions — Carbapenems; Antifungal Agents; avibactam, ceftazidime drug combination; Aztreonam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Carbapenems — First-line empirical agent for febrile neutropenia complicating hematologic malignancies: carbapenem.
Drug: Anti-Gram-positive agent — Escalation to a carbapenem plus an anti-Gram-positive agent (vancomycin or linezolid) is instituted if no defervescence occurs after 48h of first-line therapy; this combination is maintained for 3 days before further escalation in febrile-neutropenia patients with underlying hematologic malignancies.
Drug: Antifungal agent — If combination therapy with a carbapenem plus an anti-Gram-positive agent (vancomycin or linezolid) remains ineffective after 72 h, empirical antifungal coverage is added while continuing antibacterial therapy for an additional 7 days; failure to defervesce thereafter mandates further therapeutic escalation in febrile-neutropenic patients with hematologic malignancies.
Drug: Ceftazidime-avibactam + Aztreonam — If the combination of a carbapenem and an anti-Gram-positive agent (vancomycin or linezolid) fails to achieve defervescence after 3 days of treatment, an antifungal agent is added while continuing the original antibacterial regimen for an additional 7 days. Should fever persist or recur with uncontrolled infection-related parameters after 12-14 days of empirical anti-infective therapy, the carbapenem/anti-Gram-positive combination is discontinued. Therapy is then switched to ceftazidime-avibactam plus aztreonam to cover multidrug-resistant pathogens, while concurrently maintaining antifungal treatment. This escalation strategy is indicated for febrile neutropenic patients with underlying hematologic malignancies.

SUMMARY:
This single-arm, open-label clinical study evaluates the efficacy and safety of a standardized empirical anti-infective escalation protocol for patients with hematological malignancies complicated by febrile neutropenia. The treatment algorithm follows a sequential strategy: initial carbapenem monotherapy (2 days) → if ineffective, combination with vancomycin/linezolid (3 days) → if no response, escalation to antifungal therapy (7 days). For patients demonstrating persistent or recurrent fever with uncontrolled infection parameters after 12-14 days of prior empirical anti-infective therapy, switching to ceftazidime-avibactam combined with aztreonam is implemented. Therapeutic efficacy is assessed through comprehensive evaluation of clinical manifestations, inflammatory biomarkers, radiographic imaging, and microbiological findings. Comprehensive safety surveillance includes continuous monitoring of adverse events and all-cause mortality throughout the treatment course.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, observational clinical investigation focusing on patients with hematological malignancies complicated by febrile neutropenia. It aims to evaluate the overall efficacy and safety of a standardized empirical anti-infective treatment algorithm. The protocol employs a unified step-up therapeutic strategy: initial empirical administration of a carbapenem antibiotic (for 2 days); if ineffective, combination with an anti-Gram-positive agent (e.g., vancomycin or linezolid) (for 3 days); if there is still no response, initiation of antifungal therapy (for 7 days); For patients exhibiting persistent or recurrent fever with uncontrolled infection-related parameters after 12-14 days of prior empirical anti-infective therapy, an empirical multidrug-resistant regimen consisting of ceftazidime-avibactam combined with aztreonam is considered. The treatment duration will be adjusted based on neutrophil recovery and febrile status. The study will assess overall efficacy through a comprehensive evaluation of clinical symptoms and signs, inflammatory biomarkers (e.g., C-reactive protein, procalcitonin), radiographic findings, and microbiological results. Safety monitoring will include continuous surveillance of adverse events (AEs) and all-cause mortality throughout the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Documented haematological malignancy: acute leukaemia, severe aplastic anaemia, lymphoma, or multiple myeloma.
* Neutropenia: absolute neutrophil count (ANC) < 0.5 × 10⁹/L, or ANC anticipated to fall below this threshold within 48 h; severe neutropenia defined as ANC < 0.1 × 10⁹/L.
* Fever: single oral temperature ≥ 38.3 °C (axillary ≥ 38.0 °C), or oral temperature ≥ 38.0 °C (axillary ≥ 37.7 °C) sustained for > 1 h.
* Eastern Cooperative Oncology Group performance status (ECOG-PS) 0-2.
* Planned or current empirical use of ceftazidime-avibactam (CAZ-AVI) for febrile neutropenia.

Exclusion Criteria:

* Drug-related fever or fever attributable to rheumatic/autoimmune disease.
* Concomitant intracranial haemorrhage.
* Pregnancy, lactation, or intention to become pregnant.
* Psychiatric disorder or any condition precluding protocol compliance.
* Life-threatening arrhythmia or QTc > 500 ms on electrocardiography.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This single-arm, open-label, observational study will enrol adult patients with haematological malignancies who develop febrile neutropenia and are scheduled to receive empirical ceftazidime-avibactam. Eligible participants are aged 18-75 years with acute leukaemia, severe aplastic anaemia, lymphoma or multiple myeloma, an absolute neutrophil count < 0.5 × 10⁹/L (or expected to fall below this within 48 h), fever ≥ 38.3 °C, ECOG performance status 0-2, and no contraindications such as drug fever, intracranial haemorrhage, pregnancy, or QTc > 500 ms. The cohort will reflect the real-world haematology ward population at high risk for multidrug-resistant Gram-negative infections.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Symptom Resolution Rate by Patient-Reported Temperature Diary | two days
  Proportion of patients achieving defervescence (oral temperature < 38 °C sustained for ≥ 8 h) AND absence of infection-related symptoms recorded in a validated patient diary within 48 h after starting empirical therapy.
C-Reactive Protein Serum Concentration Change (mg/L) | two days
  Absolute decrease from baseline in high-sensitivity CRP measured by immunoturbidimetric assay at 48 h.
Procalcitonin Plasma Concentration Change (ng/mL) | Two days
  Absolute decrease from baseline in PCT measured by electrochemiluminescence immunoassay at 48 h.
Pulmonary Infiltrate Resolution on CT or Chest X-ray | Two weeks
  Proportion of patients with ≥ 50 % reduction in the longest diameter of any lung infiltrate compared with baseline scan.
Pathogen Positivity Rate in Blood or Sterile-Site Cultures | one week
  Cumulative proportion of patients with clinically relevant bacteria or fungi isolated from blood or other normally sterile sites processed by automated BACTEC™ culture system.
Physical Sign Resolution Score by Clinician Examination | two days
  Proportion of patients in whom predefined signs (erythema, tenderness, exudate, etc.) disappear or improve by ≥ 50 % on a 4-point clinician-graded scale.

SECONDARY OUTCOMES:
First-Line Carbapenem Clinical Success Rate | three days
  Proportion achieving defervescence AND ≥ 50 % CRP decrease at 72 h on carbapenem monotherapy.
Carbapenem Plus Anti-Gram-Positive Agent Clinical Success Rate | three days
  Proportion achieving defervescence AND ≥ 50 % CRP decrease at 72 h after adding vancomycin or linezolid.
Antifungal Therapy Biomarker Response Rate | three days
  Proportion with ≥ 50 % reduction in serum galactomannan (Platelia™ ELISA) or β-D-glucan (Fungitell™) at 72 h post-antifungal initiation.
CRE/MDR-GNB Eradication Rate After CAZ-AVI Plus Aztreonam | three days
  Proportion of patients with documented CRE/MDR-GNB whose follow-up blood or sterile-site culture becomes negative within 72 h of starting ceftazidime-avibactam plus aztreonam.
Incidence of Adverse Events Assessed by CTCAE v5.0 (Entire Course) | From first antimicrobial dose to 30 days post-therapy
  Number and grade of drug-related cardiac, hepatic, renal, or allergic adverse events captured through CTCAE v5.0 forms.
All-Cause Mortality Rate | 30 days
  Proportion of participants who die from any cause within 30 days after enrolment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China